CLINICAL TRIAL: NCT01561053
Title: A Multicenter, Randomized, Controlled Study To Evaluate The Efficacy and Safety of Short-Term Plasma Exchange Followed by Long-Term Plasmapheresis With Infusion of Human Albumin Combined With Intravenous Immunoglobulin In Patients With Mild-Moderate Alzheimer's Disease
Brief Title: A Study to Evaluate Albumin and Immunoglobulin in Alzheimer's Disease
Acronym: AMBAR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Instituto Grifols, S.A. (Industry)
Collaborators: Grifols Biologicals, LLC (Industry)
Responsible Party: Sponsor
Organization: Grifols Biologicals, LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IG1002
Record Dates: First submitted 2012-03-16; First posted 2012-03-22 (Estimated); Results first posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; Amyloid Beta (AB) peptide; Albumin; Intravenous immunoglobulin; IVIG
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid | interventions — zidovudine 5'-monophosphate-mannose-albumin conjugate; galactosamine-conjugated serum albumin-conjugated-(rhodamine X)20; Immunoglobulins; gamma-Globulins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- High Albumin + Immunoglobulin (Experimental): Therapeutic plasma exchange with albumin 5% (intensive treatment period) + Low volume plasma exchange with high dose of albumin 20% or immunoglobulin 5% (maintenance treatment period)
  Interventions: Biological: Albumin 5%; Biological: Albumin 20%; Biological: Immunoglobulin
- Low Albumin + Immunoglobulin (Experimental): Therapeutic plasma exchange with albumin 5% (intensive treatment period) + Low volume plasma exchange with low dose of albumin 20% or immunoglobulin 5% (maintenance treatment period)
  Interventions: Biological: Albumin 5%; Biological: Albumin 20%; Biological: Immunoglobulin
- Low Albumin (Experimental): Therapeutic plasma exchange with albumin 5% (intensive treatment period) + Low volume plasma exchange with low dose of albumin 20% (maintenance treatment period)
  Interventions: Biological: Albumin 5%; Biological: Albumin 20%
- Control (sham) group (No Intervention): Simulated plasma exchange procedure

INTERVENTIONS:
Biological: Albumin 5% — Therapeutic plasma exchange with human albumin 5%
  Other Names: Albutein® 5%; Human Albumin Grifols 5%
  Arms: High Albumin + Immunoglobulin; Low Albumin; Low Albumin + Immunoglobulin
Biological: Albumin 20% — Low volume plasma exchange with human albumin 5%
  Other Names: Albutein® 20%; Human Albumin Grifols 20%
  Arms: High Albumin + Immunoglobulin; Low Albumin; Low Albumin + Immunoglobulin
Biological: Immunoglobulin — Intravenous human immunoglobulin 5%
  Other Names: Flebogamma® 5% DIF
  Arms: High Albumin + Immunoglobulin; Low Albumin + Immunoglobulin

SUMMARY:
The purpose of this study is to evaluate the changes in the cognitive, functional, behavioral and global domains based on the different applicable psychometric batteries and scales.

DETAILED DESCRIPTION:
A clinical trial comprised of 350 subjects with probable mild to moderate Alzheimer's Disease (AD) will be conducted primarily to determine whether plasmapheresis with infusion of human albumin combined with intravenous immunoglobulin (IVIG) is able to modify patient's cognitive, functional, behavioral and global domains. There will be 3 treatment groups and 1 control group. The subjects will be randomized in a 1:1:1:1 proportion.

ELIGIBILITY:
Main Inclusion Criteria:

1. Males or females between 55-85 years of age at the time of signing of the informed consent document.
2. A diagnosis of Alzheimer's disease (NINCDS-ADRDA criterion), and mini-mental status examination (MMSE) score between >/=18 and </=26.
3. Current stable treatment with acetylcholine esterase inhibitors (AChEIs) and/or memantine for the previous three months.
4. The patient and a close relative or the legal representative must read the patient information sheet, agree to participation in the trial, and then sign the informed consent document (the patient personally and the close relative/legal representative).
5. The patient must be able to follow the study protocol, receive the treatment in the established time period, and continue during the follow-up interval.
6. A brain computed axial tomography (CAT) or magnetic resonance imaging (MRI) study, obtained in the 12 months prior to recruitment, showing the absence of cerebrovascular disease, should be available. Nevertheless, it is mandatory to use the MRI obtained during the screening period to rule out any cerebrovascular disease.
7. A stable care taker must be available, and must attend the patient study visits.

Main Exclusion Criteria:

1. Any contraindication for plasma exchange due to behavioral disorders or abnormal coagulation parameters, such as for example:

   * Hypocalcemia (Ca++ < 8.7 mg/dL)
   * Thrombocytopenia (<100,000/µL)
   * Fibrinogen <1.5 g/L
   * Prothrombin time (Quick) p<60% versus control (international normalized ratio (INR) >1.5)
   * Beta-blocker treatment and bradycardia <55/min
   * Treatment with angiotension-converting enzyme inhibitors (ACEIs) (increased risk of allergic reactions)
2. Hemoglobin < 10 g/dL
3. Difficult venous access precluding plasma exchange.
4. A history of frequent adverse reactions (serious or otherwise) to blood products.
5. Hypersensitivity to albumin or allergies to any of the components of Albutein.
6. History of immunoglobulin A (IgA) deficiency.
7. Known allergies to Flebogamma DIF components such as sorbitol.
8. History of thromboembolic complications of intravenous immunoglobulins.
9. Plasma creatinine > 2 mg/dl.
10. Uncontrolled high blood pressure (systolic blood pressure of 160 mmHg or higher and/or diastolic blood pressure of 100 mmHg or higher despite treatment during the last 3 months).
11. Liver cirrhosis or any liver problem with glutamic pyruvic transaminase (GPT) > 2.5 x upper limit of normal (ULN), or bilirubin > 2 mg/dL.
12. Heart diseases, as evidenced by myocardial infarction, severe or unstable angina, or heart failure (New York Association Class II, III or IV) in the past 12 months.
13. Participation in other clinical trials, or the receipt of any other investigational drug in the three months prior to the start of the study.
14. Any condition complicating adherence to the study protocol (illness with less than one year of expected survival, known drug or alcohol abuse, etc.).
15. Pregnant or nursing women or women not using effective contraceptive methods for at least one month after plasma exchange.
16. Fewer than six years of education (exclusion criteria under medical criterion).
17. Less than three months with stable treatment for behavioral disorders or insomnia.
18. Patients being treated with anticoagulants or antiplatelet therapy (antiaggregants) should not be recruited in the study.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2012-04-19 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2018-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merce Boada Rovira, MD, PhD, Principal Investigator — Fundació ACE. Barcelona. Spain; Antonio Páez, MD, Study Chair — Instituto Grifols, S.A.; Laura Núñez, BSc, Study Director — Instituto Grifols, S.A.
Locations (40):
- United States (22):
  - Northern California Research, Sacramento, California
  - Mountain View Clinical Research, Inc, Denver, Colorado
  - Howard University, Washington D.C., District of Columbia
  - Bradenton Research Center, Inc., Bradenton, Florida
  - Quantum Laboratories, Deerfield Beach, Florida
  - Galiz Research, LLC, Hialeah, Florida
  - Largo Medical Center, Largo, Florida
  - L&L Research Choices, Inc, Miami, Florida
  - Allied Biomedical Research Institute, Miami, Florida
  - Miami Dade Medical Research Institute, LLC, Miami, Florida
  - Neurology Associates of Osmond Beach, Ormond Beach, Florida
  - PharmaSeek LLC (DMI Research), Pinellas Park, Florida
  - iResearch Atlanta, LLC, Decatur, Georgia
  - RTR Medical Group, Savannah, Georgia
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - The NeuroCognitive Institute, Mount Arlington, New Jersey
  - Mid-Atlantic Geriatric/ARC, Paterson, New Jersey
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Neurology Specialists Inc, Dayton, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Roper St. Francis Healthcare, Charleston, South Carolina
  - Wesley Neurology Clinic, Cordova, Tennessee
- Spain (18):
  - Hospital General de Elche, Elche, Alicante
  - Hospital Universitario del Vinalopó, Elche, Alicante
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Hospital Universitari Mútua de Terrassa, Terrassa, Barcelona
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife, Canary Islands
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Fundació ACE, Barcelona
  - Hospital Vall d'Hebrón, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Parc Hospitalari Martí i Julià, Girona
  - Hospital Universitari de Santa Maria, Lleida
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Viamed Montecanal, Zaragoza

REFERENCES:
- [Derived] Podger L, Stewart WF, Serrano D, Lipton RB, Gomez-Ulloa D, Ayasse ND, Barnes FB, Davis EA, Runken MC. Application of a Novel Endpoint Staging Framework: Proof of Concept in the AMBAR Study. J Alzheimers Dis. 2024;98(3):1079-1094. doi: 10.3233/JAD-231197. PMID 38489186
- [Derived] Cuberas-Borros G, Roca I, Castell-Conesa J, Nunez L, Boada M, Lopez OL, Grifols C, Barcelo M, Pareto D, Paez A. Neuroimaging analyses from a randomized, controlled study to evaluate plasma exchange with albumin replacement in mild-to-moderate Alzheimer's disease: additional results from the AMBAR study. Eur J Nucl Med Mol Imaging. 2022 Nov;49(13):4589-4600. doi: 10.1007/s00259-022-05915-5. Epub 2022 Jul 22. PMID 35867135

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Albumin + Immunoglobulin | Low Albumin + Immunoglobulin | Low Albumin | Control (Sham) Group
Started | 86 | 92 | 82 | 87
Patients With Baseline MMSE:18-21 | 47 | 40 | 47 | 42
Patients With Baseline MMSE:22-26 | 39 | 52 | 35 | 45
Randomized Not Treated | 8 | 6 | 4 | 7
Evaluable Subjects | 78 | 86 | 78 | 80
Completed | 51 | 56 | 61 | 64
Not Completed | 35 | 36 | 21 | 23

BASELINE CHARACTERISTICS:
Population: 322 evaluable subjects from analysis population were defined as the overall study population (N = 347) without 25 randomized no treated subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | High Albumin + Immunoglobulin | Low Albumin + Immunoglobulin | Low Albumin | Control (Sham) Group | Total
Number analyzed (Participants) | 78 | 86 | 78 | 80 | 322
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 17 | 26 | 29 | 94
  >=65 years | 56 | 69 | 52 | 51 | 228
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.54 (7.895) | 69.47 (6.924) | 68.47 (7.476) | 68.44 (8.378) | 68.99 (7.655)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 48 | 43 | 36 | 174
  Male | 31 | 38 | 35 | 44 | 148
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Baseline Mini-Mental State Examination total score [Mean (Standard Deviation); unit: units on a scale] — Mini-Mental State Examination (MMSE) is a widely used brief 30-point questionnaire test of cognitive function among the elderly; it includes tests of orientation, registration, attention and calculation, memory (recall, naming and repetition), language (comprehension, reading and writing) and visual-spatial skills. The score ranges from 0 to 30 and is obtained by summing the points corresponding to each answer. Lower score indicates more impaired cognition.
  units on a scale | 21.41 (2.616) | 22.09 (2.633) | 21.24 (2.408) | 21.69 (2.559) | 21.62 (2.566)

OUTCOME MEASURES:

1. Primary Outcome: Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog) Total Score (Changes From Baseline to 14 Months)
Description: ADAS-Cog total score as a change from baseline to 14 months
  The ADAS-Cog Scale is a questionnaire that assesses cognitive performance in 12 different domains. The domains are: word recall, commands, constructional praxis, delayed word-recall task, naming objects/figures, ideational praxis, orientation, word recognition, remembering test instructions, comprehension, word finding difficulty, and spoken language ability. The total score ranges from 0-80 where a higher score indicates more cognitive impairment.
Time Frame: Baseline and 14 months
Population: Evaluable population with ADAS-Cog measurement at 14 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- All Treated: All patients Treatment groups 1, 2 and 3 combined
Arm/Group | High Albumin + Immunoglobulin | Low Albumin + Immunoglobulin | Low Albumin | Control (Sham) Group | All Treated
Number analyzed (Participants) | 50 | 57 | 61 | 64 | 168
units on a scale | 0.8 (1.28) | 0.8 (1.09) | 1.5 (1.02) | 3.2 (0.95) | 1.0 (0.64)

2. Primary Outcome: Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) Total Score (Changes From Baseline to 14 Months)
Description: ADCS-ADL total score as a change from baseline to 14 months
  The ADCS-ADL comprises 23 questions covering a wide array of activities of daily living. Many of the activities begin with an assessment of whether that activity is relevant and then, if yes, follow with an assessment of the difficulty. The total score over all activities ranges from 0-78 where a higher score indicates more autonomy (better outcome).
Time Frame: Baseline and 14 Months
Population: Evaluable population with ADCS-ADL measurement at 14 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | High Albumin + Immunoglobulin | Low Albumin + Immunoglobulin | Low Albumin | Control (Sham) Group | All Treated
Number analyzed (Participants) | 51 | 57 | 61 | 64 | 169
units on a scale | -3.5 (1.80) | -2.0 (1.03) | -3.9 (1.24) | -6.7 (1.50) | -3.2 (0.78)

3. Other Pre Specified Outcome: ADAS-Cog Total Score (Changes From Baseline to 14 Months) in Patients With Baseline MMSE:22-26
Description: ADAS-Cog total score as a change from baseline to 14 months in patients with baseline Mini-Mental State Examination (MMSE):22-26
  The ADAS-Cog Scale is a questionnaire that assesses cognitive performance in 12 different domains. The domains are: word recall, commands, constructional praxis, delayed word-recall task, naming objects/figures, ideational praxis, orientation, word recognition, remembering test instructions, comprehension, word finding difficulty, and spoken language ability. The total score ranges from 0-80 where a higher score indicates more cognitive impairment.
Time Frame: Baseline and 14 months
Population: Evaluable population with baseline MMSE:22-26 and with ADAS-Cog measurement at 14 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | High Albumin + Immunoglobulin | Low Albumin + Immunoglobulin | Low Albumin | Control (Sham) Group | All Treated
Number analyzed (Participants) | 23 | 37 | 25 | 38 | 85
units on a scale | -0.9 (1.51) | -0.3 (1.04) | -0.6 (1.12) | 0.6 (1.12) | -0.6 (0.68)

4. Other Pre Specified Outcome: ADCS-ADL Total Score (Changes From Baseline to 14 Months) in Patients With Baseline MMSE:22-26
Description: ADCS-ADL total score as a change from baseline to 14 months in patients with baseline Mini-Mental State Examination (MMSE):22-26
  The ADCS-ADL comprises 23 questions covering a wide array of activities of daily living. Many of the activities begin with an assessment of whether that activity is relevant and then, if yes, follow with an assessment of the difficulty. The total score over all activities ranges from 0-78 where a higher score indicates more autonomy (better outcome).
Time Frame: Baseline and 14 months
Population: Evaluable population with baseline MMSE:22-26 and with ADCS-ADL measurement at 14 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | High Albumin + Immunoglobulin | Low Albumin + Immunoglobulin | Low Albumin | Control (Sham) Group | All Treated
Number analyzed (Participants) | 23 | 37 | 25 | 38 | 85
units on a scale | -2.4 (1.68) | 0.8 (0.98) | -0.9 (1.43) | -1.3 (1.29) | -0.6 (0.75)

5. Other Pre Specified Outcome: ADAS-Cog Total Score (Changes From Baseline to 14 Months) in Patients With Baseline MMSE:18-21
Description: ADAS-Cog score as a change from baseline to 14 months in patients with baseline Mini-Mental State Examination (MMSE):18-21
  The ADAS-Cog Scale is a questionnaire that assesses cognitive performance in 12 different domains. The domains are: word recall, commands, constructional praxis, delayed word-recall task, naming objects/figures, ideational praxis, orientation, word recognition, remembering test instructions, comprehension, word finding difficulty, and spoken language ability. The total score ranges from 0-80 where a higher score indicates more cognitive impairment
Time Frame: Baseline and 14 months
Population: Evaluable population with baseline MMSE:18-21 and with ADAS-Cog measurement at 14 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | High Albumin + Immunoglobulin | Low Albumin + Immunoglobulin | Low Albumin | Control (Sham) Group | All Treated
Number analyzed (Participants) | 27 | 20 | 36 | 26 | 83
units on a scale | 2.4 (1.95) | 1.9 (2.44) | 3.3 (1.49) | 6.4 (1.34) | 2.6 (1.07)

6. Other Pre Specified Outcome: ADCS-ADL Total Score (Changes From Baseline to 14 Months) in Patients With Baseline MMSE:18-21
Description: ADCS-ADL total score as a change from baseline to 14 months in patients with baseline Mini-Mental State Examination (MMSE):18-21
  The ADCS-ADL comprises 23 questions covering a wide array of activities of daily living. Many of the activities begin with an assessment of whether that activity is relevant and then, if yes, follow with an assessment of the difficulty. The total score over all activities ranges from 0-78 where a higher score indicates more autonomy (better outcome).
Time Frame: Baseline and 14 months
Population: Evaluable population with baseline MMSE:18-21 and with ADCS-ADL measurement at 14 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | High Albumin + Immunoglobulin | Low Albumin + Immunoglobulin | Low Albumin | Control (Sham) Group | All Treated
Number analyzed (Participants) | 28 | 20 | 36 | 26 | 84
units on a scale | -4.5 (2.97) | -5.7 (2.11) | -6.0 (1.75) | -14.1 (2.67) | -5.5 (1.33)

ADVERSE EVENTS:
Time Frame: 14 Months
Description: 1 randomized subject in the control group was implanted by error with a real central catheter and was then transfered and treated as high albumin + immunoglobulin subject.
  Therefore, this subject was considered for evaluable population as control (control group [n=80] and high albumin + immunoglobulin group [n=78]), but moved to high albumin + immunoglobulin group for safety analysis (control group [n=79] and high albumin + immunoglobulin group [n=79]).
Arm/Group | High Albumin + Immunoglobulin | Low Albumin + Immunoglobulin | Low Albumin | Control (Sham) Group
All-Cause Mortality (participants affected / at risk) | 0/79 | 2/86 | 0/78 | 0/79
Serious Adverse Events (participants affected / at risk) | 16/79 | 19/86 | 8/78 | 8/79
Other Adverse Events (participants affected / at risk) | 67/79 | 77/86 | 72/78 | 56/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Albumin + Immunoglobulin (N=79) | Low Albumin + Immunoglobulin (N=86) | Low Albumin (N=78) | Control (Sham) Group (N=79)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Intentional medical device removal by patient (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis in device (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endocarditis staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaesthetic complication cardiac (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amyloid related imaging abnormalities (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Self injurious behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder neoplasm surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Knee operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Albumin + Immunoglobulin (N=79) | Low Albumin + Immunoglobulin (N=86) | Low Albumin (N=78) | Control (Sham) Group (N=79)
Anaemia (Blood and lymphatic system disorders) | 17 (17) | 17 (19) | 16 (20) | 4 (5)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 5 (5) | 1 (1) | 3 (3) | 1 (1)
Bradycardia (Cardiac disorders) | 4 (6) | 3 (3) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (6) | 6 (7) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (6) | 5 (8) | 8 (11) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 6 (6) | 5 (5) | 3 (3)
Catheter site erythema (General disorders) | 3 (4) | 3 (3) | 4 (6) | 0 (0)
Device connection issue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (8)
Extravasation (General disorders) | 10 (15) | 7 (13) | 7 (12) | 0 (0)
Infusion site extravasation (General disorders) | 7 (10) | 4 (6) | 2 (3) | 0 (0)
Oedema peripheral (General disorders) | 1 (2) | 0 (0) | 3 (3) | 5 (5)
Catheter site infection (Infections and infestations) | 1 (1) | 4 (5) | 4 (4) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (6) | 3 (3) | 7 (7) | 3 (5)
Respiratory tract infection (Infections and infestations) | 1 (1) | 4 (4) | 3 (3) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 1 (1) | 6 (6) | 5 (6)
Urinary tract infection (Infections and infestations) | 5 (6) | 6 (7) | 1 (1) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 3 (4) | 9 (10) | 4 (4) | 4 (4)
Vascular access complication (Injury, poisoning and procedural complications) | 6 (11) | 4 (5) | 4 (7) | 0 (0)
Blood fibrinogen decreased (Investigations) | 3 (4) | 5 (8) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 4 (4) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 18 (34) | 5 (6) | 9 (18) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (4) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 11 (12) | 12 (16) | 8 (10) | 3 (7)
Headache (Nervous system disorders) | 12 (13) | 4 (4) | 7 (9) | 14 (20)
Paraesthesia (Nervous system disorders) | 5 (12) | 1 (1) | 9 (16) | 0 (0)
Presyncope (Nervous system disorders) | 10 (14) | 14 (18) | 8 (9) | 2 (2)
Syncope (Nervous system disorders) | 4 (4) | 4 (5) | 4 (5) | 1 (1)
Anxiety (Psychiatric disorders) | 6 (11) | 2 (4) | 6 (6) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Haematoma (Vascular disorders) | 3 (3) | 5 (6) | 3 (4) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 3 (4) | 5 (7)
Hypotension (Vascular disorders) | 16 (34) | 16 (39) | 21 (43) | 1 (1)
Poor venous access (Vascular disorders) | 7 (10) | 6 (7) | 4 (6) | 0 (0)
Catheter site pain (General disorders) | 2 (2) | 0 (0) | 9 (11) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A 18-month post-study period is reserved for a joint, multi-center publication of study results. After this period, individual sites may publish results provided that the Sponsor is allowed 60 days to review any proposed publication for removal of confidential, protected, and trademarked material prior to submission with an option to delay publication up to 120 days if needed to protect its interests. The Sponsor shall retain the option to receive acknowledgment for its sponsorship of the study.

DOCUMENTS (2):
  • Study Protocol (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/53/NCT01561053/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/53/NCT01561053/SAP_001.pdf